CLINICAL TRIAL: NCT05769933
Title: Fine-scale Mapping of Brain Anatomy and Function With Combined Electroencephalography and 7T Magnetic Resonance Imaging: a Single-center Study on Healthy Participants and on Tremor, Psychosis and Epilepsy Patients
Brief Title: Bridging Gaps in the Neuroimaging Puzzle: New Ways to Image Brain Anatomy and Function in Health and Disease Using Electroencephalography and 7 Tesla Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Collaborators: Institute for Diagnostic and Interventional Neuroradiology, Inselspital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 221-FP.2333_PUZZLE; SNCTP000005245 (Other: Coordination Office for Human Research (kofam), Switzerland)
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Healthy; Epilepsy; Psychosis; Essential Tremor
Keywords: electroencephalography; magnetic resonance imaging; ultra-high field; neuroimaging
MeSH Terms: conditions — Epilepsy; Psychotic Disorders; Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy participants: Healthy volunteers with no history of neurological problems or mental disorders; normal vision or corrected-to-normal using contact lenses. Interventions: MRI and combined EEG-fMRI.
  Interventions: Device: Simultaneous EEG-fMRI at 7 Tesla; Device: Structural MRI at 7 Tesla
- Essential tremor patients: Non-hospitalized volunteers who have been diagnosed with essential tremor and are indicated for thalamic surgery. Interventions: MRI.
  Interventions: Device: Structural MRI at 7 Tesla
- Psychosis patients: Non-hospitalized volunteers who have been diagnosed with early psychosis, and clinically assessed; normal vision or corrected-to-normal using contact lenses. Interventions: MRI and combined EEG-fMRI.
  Interventions: Device: Simultaneous EEG-fMRI at 7 Tesla; Device: Structural MRI at 7 Tesla
- Healthy controls: Healthy volunteers who have been clinically assessed and determined to be suitable matched controls with respect to the psychosis group; normal vision or corrected-to-normal using contact lenses. Interventions: MRI and combined EEG-fMRI.
  Interventions: Device: Simultaneous EEG-fMRI at 7 Tesla; Device: Structural MRI at 7 Tesla
- Epilepsy patients: Non-hospitalized volunteers who have been diagnosed with epilepsy.
  Interventions: Device: Simultaneous EEG-fMRI at 7 Tesla; Device: Structural MRI at 7 Tesla

INTERVENTIONS:
Device: Simultaneous EEG-fMRI at 7 Tesla — Scalp electroencephalography (EEG) and functional magnetic resonance imaging (MRI) at 7 Tesla. These will be completely non-invasive techniques with no ionizing radiation and no injected contrasts.
  Groups: Epilepsy patients; Healthy controls; Healthy participants; Psychosis patients
Device: Structural MRI at 7 Tesla — Structural magnetic resonance imaging (MRI) at 7 Tesla. These will be completely non-invasive techniques with no ionizing radiation and no injected contrasts.

SUMMARY:
The human brain presents outstanding challenges to science and medicine. Brain function and structure span broad spatial scales (from single neurons to brain-wide networks) as well as temporal scales (from milliseconds to years). Currently, none of the tools available for studying the brain can fully capture its structure and function across these diverse scales - "the neuroimaging puzzle". This poses crucial limitations to understanding how the brain works, and how it is affected by numerous diseases.

The central goal of this project is to expand currently available tools for non-invasive human brain imaging, to bridge critical gaps in the neuroimaging puzzle. New methodologies will be developed, focused on ultra-high field magnetic resonance imaging (UHF MRI) and its combination with electroencephalography (EEG). New contrast mechanisms and technological advances enabled by UHF MRI and EEG will be explored to allow unprecedented views into the microstructure of brain regions like the thalamus, and to capture the activity of large-scale neuronal networks in the brain with high sensitivity, temporal and spatial specificity. These advances will be directly applied to address open questions in the diagnosis and treatment of essential tremor, and psychosis.

In general, improved brain imaging techniques are critical for a deeper understanding of how the brain works, and to detect and characterize diseases more effectively, thereby improving clinical management and leading to a healthier population. The non-invasive characterization and treatment of neurodegenerative diseases like tremor is particularly relevant to aging modern societies.

ELIGIBILITY:
Inclusion Criteria:

* Common to all participant groups: be 18 years old or older; be able to understand instructions; be able to provide informed consent.
* Specific to healthy participants: have no history of neurological or mental disorders; normal vision or corrected-to-normal using contact lenses.
* Specific to the patient groups: not be hospitalized; having been diagnosed with tremor, epilepsy or psychosis and invited to participate by our team's clinicians; for some groups: normal vision or corrected-to-normal using contact lenses.

Exclusion Criteria:

* Contra-indications for MRI (e.g. an implant that is not MRI-compatible), also including having claustrophobia or being pregnant.
* Inability to follow the necessary tasks of the study (e.g. unable to lie on the scanner bed).
* Having undergone brain surgeries in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers and adult patients without specific risk profiles.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Contrast-to-noise ratio between thalamic nuclei in 7T structural MRI | Day 1
Pearson correlation between thalamocortical brain regions in 7T functional MRI | Day 1
Microstate duration in EEG acquired concurrently with 7T functional MRI | Day 1

SECONDARY OUTCOMES:
Neuroimaging datasets published in fully anonymized form in suitable public data repositories | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- TIC - Translational Imaging Center, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Neuroimaging data from the study will be made publicly available in fully anonymized form.
Time Frame: With relevant publications
Access Criteria: Publicly available (anonymized)